CLINICAL TRIAL: NCT06085235
Title: An Investigation Into the Effects of Acute Exercise on Activities of Daily Living and Cognition in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Principal Investigator, Jean-Charles Lebeau, Assistant Professor of Sport and Exercise Psychology, Ball State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1141661-20
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial: exercise or video control condition
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): 15min of cycling at moderate intensity
  Interventions: Behavioral: exercise
- video control (No Intervention): watching a video on healthy living

INTERVENTIONS:
Behavioral: exercise — cycling exercise for 15min, with 5min warm up
  Arms: exercise

SUMMARY:
Research has demonstrated the positive effects of chronic exercise on cognitive functioning and performance of Activities of Daily Living (ADLs). However, minimal research exists regarding the effects of acute exercise. To address this gap in the literature, the present study investigated the effect of an acute bout of exercise on executive functions, balance, and ADLs among healthy older adults. Based on the current literature, we expected participants in the exercise group to perform better on executive function tasks and ADLs compared to participants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 60.

Exclusion Criteria:

* health complications preventing the ability to cycle on a recumbent bike and walking at moderate intensity as indicated by the health history questionnaire, taking anti-depressant medication, or having color blindness.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Executive functions | 1 week
  Stroop test. The Stroop test is a measure of executive functions, specifically the ability to inhibit a habitual response, selective attention, and shifting (Pachana et al., 2014). This test requires participants to identify the color name printed in the same ink color (e.g., BLUE printed in blue ink; congruent condition) or different ink color (e.g., BLUE printed in red ink; incongruent condition). Each stimulus word (i.e., red, green, and blue) was presented in equal proportions to minimize specific word facilitation. After nine practice trials, 72 stimuli (i.e., 2 blocks of 36) were presented to the participants using the Eprime software (Version 3.0). Participants were asked to press the key with the dot sticker corresponding to the three stimuli colors (i.e., red, blue, or green). Reaction time (RT) and accuracy were used as indices of performance.
Balance | 1 week
  Berg Balance Scale (BBS). The BBS was developed to measure balance and fall risk among older adults. This scale is comprised of 14 tasks to assess balance, such as standing with eyes closed and retrieving an object from the floor. Performance is rated on a 0 to 4 scale for each task, with "0" indicating the lowest level of function and "4" the highest level of function. Total scores of 41 to 56 indicate a low fall risk, 21 to 40 a medium fall risk, and 0 to 20 a high fall risk (Berg et al., 1992).
Activity of daily living | 1 week
  Medication task. A medication task was developed to test the participants' ability to properly complete their pill organizers. Participants read a fictional story about prescribed medications and were asked to determine the required frequency and dosage of the medications based on the prescription and the label on fake medication bottles filled with candy pills. Participants had to place the medications in a weekly pill organizer for each required day and time slot (AM and PM). Two scenarios were designed to both require a similar number of pills to be placed in the weekly container for pre and post-test. Time to complete the task and number of mistakes for each day and time slot were recorded as indices of performance. Mistakes were recorded when participants added too many or too little pills, when pills were placed in the incorrect AM/PM time slot, or when participants added the wrong type of medication on a given day.
Functional ability | 1 week
  15 feet task. The 15-feet task measures functional ability in older adults. Participants are instructed to walk for 15 feet at their own pace while their performance is timed.
Fall risk | 1 week
  Time up and go (TUG). The TUG is used to measure fall risk in the elderly population and consists of instructing the participant to stand up from a chair, walk three meters, turn around, walk back, and sit down in the chair. The participants were instructed to walk at their regular pace and performance was measured as the time required to complete the activity. A timed score of greater than 14 seconds indicated a high risk of falls (Bohannon, 2006).
Grip strength | 1 week
  Grip strength. Verbecq et al. (2017) reported that low muscle strength, as measured by hand grip strength, was associated with a history of falls in older adults To measure hand grip strength, participants were asked to squeeze the handle of a handgrip dynamometer as hard as possible with their dominant hand and the mean score of three trials was recorded.
Commitment check | 1 week
  A commitment check was developed to test participants' commitment to the tasks. Participated were asked how committed they were while performing (a) the Stroop task, (b) the medication task, (c) the BBS tasks, (d) the TUG task, and (e) the grip strength task. Each item was rated on a scale ranging from 1 (none / not at all) to 10 (very much / very well).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Lebeau, PHD, Principal Investigator — Ball State University
Locations (1):
- Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
dataset
Time Frame: available immediately, no time frame
URL: https://osf.io/y8e2r/

REFERENCES:
- Available data/document: Individual Participant Data Set — https://osf.io/y8e2r/